CLINICAL TRIAL: NCT00129350
Title: An Assessment of Patient Outcomes Following a Rehabilitation Programme for Patients Who Have Received Lung or Heart-Lung Transplant - a Randomised Controlled Trial
Brief Title: Assessment of Heart and Heart-Lung Transplant Patient Outcomes Following Pulmonary Rehabilitation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-069; 2004NU005B
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Last update posted 2005-09-07 (Estimated); Status verified 2005-08

CONDITIONS: Emphysema; Alveolitis, Fibrosing; Cystic Fibrosis; Bronchiectasis; Lung Diseases
Keywords: End Stage Fibrotic Lung Disease
MeSH Terms: conditions — Emphysema; Pulmonary Fibrosis; Cystic Fibrosis; Bronchiectasis; Lung Diseases

INTERVENTIONS:
Procedure: Pulmonary rehabilitation programme

SUMMARY:
At present, a specific community based rehabilitation programme for lung or heart-lung transplant recipients does not exist. 160 hospitals throughout the United Kingdom (UK) offer pulmonary rehabilitation programmes. The programmes operate under evidence-based guidelines as outlined by the Chartered Society of Physiotherapy. Increasing evidence shows that rehabilitation programmes help improve performance, exercise endurance, and quality of life; and reduce symptoms and demand on health-care resources. This study proposes to compare the outcomes of lung and heart-lung transplant patients attending local pulmonary rehabilitation against others receiving the Trust's current document-based programme. The study is a randomized controlled trial:

* Control Arm: Those patients randomized to the 'control' arm will receive the Trust's standard rehabilitation programme that consists of an information pack supplied upon discharge. They will then complete and undertake the following tests: Short-Form 36 (SF 36; version 2) Questionnaire, Chronic Respiratory Questionnaire (CRQ-SR), Incremental Shuttle Walk Test and Spirometry forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC). The patient will follow the information contained in the information pack and the above tests and questionnaires will be repeated 6 months post discharge.
* Experimental Arm: A patient who is randomized to the 'experimental' arm will be asked to complete the following tests upon discharge: Short-Form 36 (SF 36; version 2) Questionnaire, Chronic Respiratory Questionnaire (CRQ-SR), Incremental Shuttle Walk Test and Spirometry FEV1 and FVC. Three months post discharge, the patient will be enrolled into a local pulmonary rehabilitation programme. The programme is typically structured to last 6-12 weeks. The above tests and questionnaires will be repeated 6 months post discharge.

To measure the effectiveness of either the information pack or the rehabilitation programme the following endpoints will be subjected to analysis in both the experimental and the control group:

* Short-Form 36 Questionnaire;
* Chronic Respiratory Questionnaire;
* Incremental Shuttle Walk Test;
* Borg Scale;
* Spirometry FEV1 and FVC;
* Hospital re-admission rates and mortality rates.

The undertaking of a multidisciplinary-led programme of rehabilitation facilitates a better quality of life than a document-based rehabilitation programme in lung and or heart-lung transplant out-patients.

The aim of the study is to construct an optimal programme of rehabilitation in lung or heart-lung patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone either a lung or heart-lung transplant.
* Fit for discharge from the Transplant Unit's Intensive Care Unit.
* > 18 years of age.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients unable to understand or comprehend the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2008-02

PRIMARY OUTCOMES:
Exercise Shuttle Test (metres completed)

SECONDARY OUTCOMES:
Borg score
Quality of life: SF-36 and Chronic Respiratory Questionnaires
Spirometry
Hospital re-admission rates
Organ rejection

CONTACTS AND LOCATIONS:
Overall Officials: MARTIN CARBY, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Harefield Hospital, Harefield, United Kingdom

REFERENCES:
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853